CLINICAL TRIAL: NCT00252161
Title: Randomized Phase III Trial of Surgery Plus Neoadjuvant TS-1 and Cisplatin Compared With Surgery Alone for Type 4 and Large Type 3 Gastric Cancer: Japan Clinical Oncology Group Study (JCOG 0501)
Brief Title: A Trial of Neoadjuvant TS-1 and Cisplatin for Type 4 and Large Type 3 Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haruhiko Fukuda (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Sponsor-Investigator, Haruhiko Fukuda, JCOG Data Center, Japan Clinical Oncology Group
Organization: Japan Clinical Oncology Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG0501; C000000279 (Registry Identifier: UMIN-CTR)
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Gastric Neoplasm
Keywords: Neoadjuvant Therapy; Stomach Neoplasms; Cisplatin; S-1(combination)
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Procedure/Surgery: Gastrectomy with more than D2 dissection
  Interventions: Procedure: Gastrectomy with more than D2 dissection
- 2 (Experimental): Drug: Neoadjuvant chemotherapy(TS-1+CDDP) followed by gastrectomy
  Interventions: Drug: Neoadjuvant chemotherapy(TS-1+CDDP) followed by gastrectomy

INTERVENTIONS:
Procedure: Gastrectomy with more than D2 dissection — Gastrectomy with more than D2 dissection
  Arms: 1
Drug: Neoadjuvant chemotherapy(TS-1+CDDP) followed by gastrectomy — Neoadjuvant chemotherapy(TS-1+CDDP) followed by gastrectomy
  Arms: 2

SUMMARY:
The aim of this study is to evaluate survival benefit of TS-1 plus cisplatin as a neoadjuvant chemotherapy in gastric cancer patient with resectable type 4 (linitis plastica type) and large type 3 tumor in comparison with surgery alone.

DETAILED DESCRIPTION:
A randomized phase III study is going to started in Japan to compare TS-1 plus cisplatin as a neoadjuvant chemotherapy with surgery alone in patient with type 4 and large type 3 gastric cancer.A total of 300 patients will be accrued for this study from 35 institutions within five years. The primary endpoint is overall survival. The secondary endpoints are progression free survival (PFS), response rate, proportion of protocol achievement, proportion of curative resection, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. histologically proven adenocarcinoma of stomach
2. Borrmann type 4 or large (>=8 cm) type 3
3. no evidence of distant metastasis including liver(M0)
4. no evidence of para-aortic and/or retropancreatic lymph node metastasis(N0-2)
5. no peritoneal metastasis and negative peritoneal lavage cytology (PLS) with laparoscopic confirmation
6. no involvement of the esophagus with > 3cm
7. an age of 20-75 years
8. an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
9. no prior chemotherapy, radiotherapy for any malignancy
10. no prior surgery for gastric cancer except for endoscopic membrane resection (EMR)
11. no breeding from primary tumor or gastrointestinal stenosis
12. sufficient oral intake
13. adequate organ function
14. written informed consent

Exclusion Criteria:

1. synchronous or metachronous (within 5 years) malignancy other than carcinoma in situ
2. pregnant or breast-feeding women
3. severe mental disease
4. systemic administration of corticosteroids, flucytosine, phenytoin or warfarin
5. other severe complications such as paralytic ileus, intestinal pneumonitis, pulmonary fibrosis, or ischemic heart disease
6. myocardial infarction within six disease-free months

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2005-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
overall survival | during the study conduct

SECONDARY OUTCOMES:
progression free survival (PFS) | during the study conduct
response rate | during the study conduct
proportion of protocol achievement | during the study conduct
proportion of curative resection | during the study conduct
adverse events | during the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Mitsuru Sasako, MD, PhD, Study Chair — Hyogo Medical University
Locations (35):
- Japan (35):
  - Aichi Cancer Center Hospital, Nagoya,Chikusa-ku,Kanokoden,1-1, Aichi-ken
  - Fujita Health University, Toyoake,Kutsukake-cho,Dengakugakubo,1-98, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa,Kashiwanoha,6-5-1, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama,Horinouchi,13, Ehime
  - Gifu Municipal Hospital, Gifu,Kashima-cho,7-1, Gifu
  - Hiroshima City Hospital, Hiroshima,Naka-ku,Motomachi,7-33, Hiroshima
  - Itami City Hospital, Itami,Koyaike,1-100, Hyōgo
  - Iwate Medical University, Morioka,Uchimaru,19-1, Iwate
  - Kagoshima University,Faculty of Medicine, Kagoshima,Sakuragaoka,8-35-1, Kagoshima-ken
  - Kanagawa Cancer Center, Yokohama,Asahi-ku,Nakao,1-1-2, Kanagawa
  - Kyoto Second Red Cross Hospital, Kamigyo-ku,Kamanza-Marutamachi,355-5, Kyoto
  - Miyagi Cancer Center, Natori,Medeshima-Shiode,Nodayama,47-1, Miyagi
  - National Hospital Organization, Sendai Medical Center, Sendai,Miyagino-ku,Miyagino,2-8-8, Miyagi
  - Nagaoka Chuo General Hospital, Nagaoka,Kawasaki,2041, Niigata
  - Niigata Cancer Center Hospital, Niigata,Kawagishi-cho,2-15-3, Niigata
  - Tsubame Rosai Hospital, Tsubame,Sawatari,633, Niigata
  - Oita University Fuculty of Medicine, Oita,Hasama-machi,Oogaoka,1-1, Oita Prefecture
  - Osaka National Hospital, Osaka,Chuo-ku,Hoenzaka,2-1-14, Osaka
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka,Higashinari-ku,Nakamichi,1-3-3, Osaka
  - Kinki University School of Medicine, Osaka-Sayama,Ohno-higashi,377-2, Osaka
  - Sakai Municipal Hospital, Sakai,Minamiyasuicho,1-1-1, Osaka
  - Osaka Medical College, Takatsuki,Daigakucho,2-7, Osaka
  - Toyonaka Municipal Hospital, Toyonaka,Shibaharacho,4-14-1, Osaka
  - Saitama Cancer Center, Kita-adachi,Ina,Komuro,818, Saitama
  - National Defense Medical College, Tokorozawa,Namiki,3-2, Saitama
  - Shizuoka General Hospital, Shizuoka,Aoi-ku,Kitaando,4-27-1, Shizuoka
  - Tokyo Metropolitan Komagome Hospital, Bunkyo-ku,Honkomagome,3-18-22, Tokyo
  - Tokyo Medical and Dental University Hospital, Bunkyo-ku,Yushima,1-5-45, Tokyo
  - National Cancer Center Hospital, Chuo-ku,Tsukiji,5-1-1, Tokyo
  - Cancer Institute Hospital, Koto-ku,Ariake,3-10-6, Tokyo
  - International Medical Center of Japan, Shinjuku-ku,Toyama,1-21-1, Tokyo
  - Tokyo Metropolitan Bokutoh Hospital, Sumida-ku,Koutoubashi,4-23-15, Tokyo
  - Toyama Prefectural Central Hospital, Toyama,nishinagae,2-2-78, Toyama
  - Wakayama Medical University, School of Medicine, Wakayama,Kimiidera,811-1, Wakayama
  - Yamagata Prefectural Central Hospital, Yamagata,Aoyagi,1800, Yamagata

REFERENCES:
- See also: Related Info — http://www.jcog.jp/